CLINICAL TRIAL: NCT05374304
Title: Improving Decision Making for Older Adults With Cancer: A Feasibility Pilot Study
Brief Title: Decision Making for Older Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Mount Zion Health Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22052; 1K76AG064431 (NIH)
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Cancer
Keywords: Geriatric Oncology; Decision Making
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial (CRT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lead-In (BC/WC-GeriOnc) (Experimental): Lead-in phase oncologists will complete the BC/WC-GeriOnc communication tool training. Cancer treatment decision-making discussions will be recorded with 2 patients per oncologist and ask patients and oncologists to complete study questionnaires over one-month follow-up and one semi-structured interview about the decision-making process and communication.
  Interventions: Other: Best Case/Worst Case (BC/WC) Geriatric Oncology (GeriOnc) communication tool
- Intervention (BC/WC-GeriOnc) (Experimental): Intervention group oncologists will complete the BC/WC-GeriOnc communication tool training. Cancer treatment decision-making discussions will be recorded with 2 patients per oncologist to understand baseline oncologist practices and communication. Patients and oncologists will be asked to complete study questionnaires over a 2 month follow-up and 1 semi-structured interview. For each randomized oncologist, cancer treatment decision-making discussions will be recorded with 5 patients per oncologist. Both patients and oncologists will also be asked to complete study questionnaires over a 2 month follow-up and 1 semi-structured interview about the decision-making process and communication. Each patient will be given the option to select 1 caregiver to participate. Caregivers will be asked to complete study questionnaires and a semi-structured interview about their decision-making experience.
  Interventions: Other: Best Case/Worst Case (BC/WC) Geriatric Oncology (GeriOnc) communication tool
- Waitlist Control (No Intervention): Usual care will be provided to the patients, with optional training for the oncologists at study completion.

INTERVENTIONS:
Other: Best Case/Worst Case (BC/WC) Geriatric Oncology (GeriOnc) communication tool — The BC/WC framework guides clinicians to present a choice between two options and uses scenario planning (narrative descriptions of plausible outcomes that acknowledge uncertainty) to describe the best, worst, and most likely case for each option. Scenarios are informed by clinical judgement and knowledge of patient risk factors. These scenarios plus an accompanying graphic aid help patients formulate and express preferences and concerns about treatment burdens and outcomes. The clinician then provides a goal-concordant recommendation.
  Other Names: BC/WC GeriOnc communication tool
  Arms: Intervention (BC/WC-GeriOnc); Lead-In (BC/WC-GeriOnc)

SUMMARY:
This is a minimal risk, pilot cluster randomized controlled trial (CRT) to determine the feasibility and acceptability of training medical oncologists to use the Best Case/Worst Case-Geriatric Oncology (BC/WC-GeriOnc) communication tool in clinical practice with older adults with cancer.

DETAILED DESCRIPTION:
Primary Objective:

I. To assess the feasibility of study procedures and using the BC/WC-GeriOnc communication tool in medical oncology with older adults with cancer.

Secondary Objectives

I. To evaluate the acceptability and appropriateness of using the BC/WC-GeriOnc communication tool.

II. To evaluate BC/WC-GeriOnc intervention fidelity and adherence by oncologists .

Exploratory Objectives:

I. To assess shared decision making and qualitatively compare cancer decision-making discussions led by oncologists randomized to the BC/WC-GeriOnc intervention versus control.

II. To determine the variability in physician-patient communication and decision-making outcomes in the intervention and control groups III. To characterize cancer care decisions and health care utilization in the intervention and control groups.

During the lead-in phase, 2 medical oncologists and 4 participants will be enrolled. During the CRT, 7 medical oncologists, 49 patients, and up to 42 caregivers will be enrolled.

Oncologists will then be randomized 1:1 to the BC/WC-GeriOnc intervention arm or waitlist control with optional BC/WC-GeriOnc training after study completion. For each randomized oncologist, the investigators will record cancer treatment decision-making discussions with 5 patients per oncologist and ask participants and oncologists to complete study questionnaires over two-month follow-up and one semi-structured interview about the decision-making process and communication.

Each participant in the pilot CRT phase will be given the option to select one caregiver to participate as well. Caregivers will be asked to complete study questionnaires and a semi-structured interview about their decision-making experience.

ELIGIBILITY:
Inclusion Criteria for Oncologists:

1. Independently practicing medical oncology physician (non-ACGME oncology fellows who practice independently are eligible).
2. Annually care for at least 10 patients age >=65 years with solid tumor malignancies in the outpatient setting (this criterion will be confirmed by oncologist report).
3. Willing to complete the two-hour intervention training.
4. At the time of enrollment, plans to continue outpatient practice at a University of California, San Francisco (UCSF) Helen Diller Family Comprehensive Cancer Center (HDFCCC) affiliated site for the duration of the pilot study.

Inclusion Criteria for Patients:

1. Age >= 65 years.
2. Diagnosed with a solid tumor malignancy of any stage.
3. 3. Upcoming decision-making discussion (in-person or via video conferencing) with a participating medical oncologist.
4. Able to read, write, and understand English.
5. Able to understand and provide written, informed consent. Adequate decisional capacity to consent for this study will be determined using the UCSF Decision-Making Capacity Assessment Tool. Patients with mild cognitive impairment who have adequate decisional capacity to consent for this study will be included.

There are no performance status, organ function, or comorbidity eligibility criteria for this study.

During the CRT phase, patients will be given the option to select a caregiver to participate in the study (not required). Caregivers cannot participate without an enrolled patient. Caregivers may be a family member, partner, or friend of the participating patient.

Inclusion Criteria for Caregivers:

1. Age >=18 years.
2. Must plan to be present during the medical oncology decision-making discussion and follow-up visits within the first 3 months.
3. Able to read, write, and understand English.
4. Able to understand and provide written, informed consent.

Exclusion Criteria:

Exclusion Criteria for Oncologists:

1. Medical oncologists who practice solely in the inpatient setting are not eligible.

Exclusion Criteria for Patients:

1. Plan for UCSF second opinion evaluation only. Patients are eligible if they plan to transfer care to UCSF at the time of enrollment.
2. Planned decision-making discussion via phone only (without video).
3. Patients participating in another cancer communication/decision support intervention study with their medical oncologist.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | 1 day
  Proportion of eligible patients who enroll in the study. An enrollment rate >=50% will be used to determine overall feasibility, which was selected based on decreased enrollment observed in studies of older adults with cancer during the ongoing 2019 novel coronavirus (COVID-19) pandemic.
Retention rate | 3 months
  Proportion of oncologists, participants, and caregivers who complete the study. A completion rate of >=75% study completion excluding drop out due to death will be used to determine overall feasibility.
Duration of audio-recorded decision-making discussions | Within 2 weeks after cancer care decision is made for each participating patient
  The duration of audio-recorded decision-making discussions in the intervention group will be compared with the duration in the control group. The investigators will compare the duration of the overall patient visit, the decision-making discussion portion of the patient visit, and the decision-making discussion portion of the patient visit plus any subsequent follow-up discussions until the decision is made.
Feasibility of Intervention Measure (Lead-In and BC/WC-GeriOnc Intervention Groups Only) | Within 2 weeks after cancer care decision is made for each participating patient
  Oncologists will complete the Feasibility of Intervention Measure, which includes 4 items with responses rated on a 5-point Likert scale from completely disagree to completely agree. The measure is scored by calculating the mean of the responses with a higher score indicating greater feasibility.
Qualitative oncologist-reported feasibility (Lead-In and BC/WC-GeriOnc Intervention Groups Only) | Completed once at the end of study participation (approximately 18 months)
  Oncologists will participate in one semi-structured interview at study completion to learn about their perspectives on intervention feasibility.

SECONDARY OUTCOMES:
Practitioner Opinion Survey (Lead-In and BC/WC-GeriOnc Intervention Groups Only) | Completed once at the end of study participation (approximately 18 months)
  Oncologists will complete the Practitioner Opinion Survey, which includes 15 items to assess physician perspectives on using a decision aid including ease of use and benefits compared with their usual approach. The investigator will modify the survey to refer to BC/WC-GeriOnc as the intervention.
Acceptability of Intervention Measure (Lead-In and BC/WC-GeriOnc Intervention Groups Only) | Within 2 weeks after cancer care decision is made for each participating patient
  Oncologists will complete the Acceptability of Intervention Measure, which includes 4 items with responses rated on a 5-point Likert scale from completely disagree to completely agree. The measure is scored by calculating the mean of the responses with a higher score indicating greater acceptability.
Intervention Appropriateness Measure (Lead-In and BC/WC-GeriOnc Intervention Groups Only) | Within 2 weeks after cancer care decision is made for each participating patient
  Oncologists will complete the Intervention Appropriateness Measure, which includes 4 items with responses rated on a 5-point Likert scale from completely disagree to completely agree. The measure is scored by calculating the mean of the responses with a higher score indicating greater appropriateness.
BC/WC-GeriOnc Intervention Fidelity (Lead-In and BC/WC-GeriOnc Intervention Groups Only) | Within 2 weeks after cancer care decision is made for each participating patient
  The BC/WC-GeriOnc Communication Tool Skills Checklist will used to assess intervention fidelity by evaluating audio-recordings and graphic aids after each use of BC/WC-GeriOnc. The BC/WC-GeriOnc Communication Tool Skills Checklist was adapted from the original 15-item checklist for the BC/WC communication tool. This checklist includes essential elements of the intervention and will be used to evaluate oncologist proficiency at the end of intervention training and to assess fidelity to the intervention during the study.
BC/WC-GeriOnc Intervention Adherence (Lead-In and BC/WC-GeriOnc Intervention Groups Only) | Within 2 weeks after cancer care decision is made for each participating patient
  Proportion of study visits with participating patients during which oncologists use the BC/WC-GeriOnc communication tool.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Debouer, MD, MA, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - San Francisco Veterans Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT05374304/ICF_000.pdf